CLINICAL TRIAL: NCT01618448
Title: A Multicenter, Double-blind, Randomized, Placebo-Controlled Study to Evaluate the Efficacy and Safety of Tolvaptan in the Treatment of Cardiac-Induced Edema in Patients With Heart Failure
Brief Title: Efficacy and Safety of Tolvaptan in the Treatment of Cardiac-Induced Edema in Patients With Heart Failure
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Taiwan Otsuka Pharm. Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 156-TWA-1101
Record Dates: First submitted 2012-06-05; First posted 2012-06-13 (Estimated); Last update posted 2015-06-02 (Estimated); Status verified 2013-01

CONDITIONS: Cardiac-induced Edema
MeSH Terms: conditions — Edema, Cardiac | interventions — Tolvaptan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Experimental): Placebo once daily
  Interventions: Drug: Placebo
- Tolvaptan (Experimental): Tolvaptan 15mg once daily
  Interventions: Drug: Tolvaptan

INTERVENTIONS:
Drug: Tolvaptan — Tolvaptan 15mg once daily
  Other Names: Samsca
  Arms: Tolvaptan
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
A Multicenter, Double-blind, Randomized, Placebo-Controlled Study to Evaluate the Efficacy and Safety of Tolvaptan in the Treatment of Cardiac-Induced Edema in Patients with Heart Failure

DETAILED DESCRIPTION:
Interventional, phase III, 2-arm parallel group, placebo-controlled, multicenter, randomized 1:1, double-blind study, comparing Tolvaptan and placebo in hospitalized HF patients with signs or symptoms of congestion at the time of randomization in spite of standard therapy.This study intends to demonstrate that a repeated 4-day treatment with Tolvaptan in addition to standard of care (SOC) is superior to SOC alone for the treatment of clinical relevant cardiac-induced volume retention parameters in patients hospitalized for worsening HF initially treated with conventional therapy including diuretics.

ELIGIBILITY:
Inclusion Criteria:

2. Patients with history of chronic HF hospitalized primarily for worsening HF with signs or symptoms of volume congestion in spite of standard therapy 3. Patient should have HF symptoms at rest or minimal exertion and signs of congestion (lower limb edema, jugular venous distention, or pulmonary congestion due to extracellular volume expansion) at time of randomization c. Anti-aldosterone drugs: Spironolactone, Triamterene 4. Patients undergoing any of the following diuretic therapies:

* A loop diuretic at a daily dosage equivalent to 40 mg or more of furosemide
* Concomitant administration of a loop diuretic and a thiazide diuretic (at any doses)
* Concomitant administration of a loop diuretic and an anti-aldosterone drug (at any doses)

Note: The allowable types and dosages of the concomitantly administered diuretics are specified as follows:

1. Loop diuretics equivalent to 40 mg of furosemide:

   Bumetanide: 1 mg, Piretanide: 6 mg, Azosemide: 60 mg, Torasemide: 8 mg
2. Thiazide diuretics: Hydrochlorothiazide, Trichloromethiazide, Benzyl hydrochlorothiazide, Chlortalidone, Mefruside 5. Patients who had been taking an orally administered diuretic without any change in dose or mode of administration during Observation period 6. Patients whose body weight variation was within 1.0 kg during the 2 days prior start of treatment 7. Patients able to accomplish with study procedures from Screening period to Post-study follow-up 8. Patients capable of giving informed consent to participate in the study of their own free will.

Exclusion Criteria:

1. Cardiac surgery within 60 days of enrollment
2. Patients with an assisted cardiac mechanical device
3. Patients receiving CRT (Cardiac Resynchronization Therapy) within 60 days of enrollment.
4. Patients with active or significant complications or symptoms as follow:

   * Suspected decrease in circulatory blood flow
   * Refractory end-stage HF (patients considered to require mechanical circulatory support, continuous intravenous positive inotropic therapy, referral of cardiac transplantation, or hospice care)
   * Cardiac valvular disease with significant heart valve stenosis
   * Sustained ventricular tachycardia or ventricular fibrillation within 30 days prior to screening examination
   * Acute myocardial infarction within 30 days prior to screening examination
   * Cerebrovascular disorders within 6 months prior to screening examination (other than asymptomatic cerebral infarction)
   * Patients with a definite diagnosis of active myocarditis or amyloid cardiomyopathy
   * Poorly controlled Diabetes Mellitus (HbAlc 10%)
   * Anuria (urinary output less than 100 ml per day)
   * History of Hyperthyroidism
   * Urination impaired due to urinary tract stricture, urinary calculus, tumor in urinary tract, or other cause
   * Hemofiltration or dialysis
   * Patients unable to sense thirst, inappropriately respond to thirst or those who have impaired oral fluid intake.
5. Patients with a history of hypersensitivity or idiosyncratic reaction to benzazepine derivatives such as mozavaptan hydrochloride or benazepril hydrochloride
6. Patients who are severely obese (BMI exceeding 35 kg/m2)
7. Patients with systolic blood pressure in the decubitus position below 90 mmHg
8. Patients with any of following abnormal laboratory values:

   Total bilirubin exceeding 3.0 mg/dL, hemoglobin of less than 9 g/dL, serum creatinine exceeding 3.0 mg/dL, serum sodium exceeding 147 mEq/L, or serum potassium exceeding 5.5 mEq/L
9. Female patients who are pregnant, possibly pregnant, or lactating, or who plan to become pregnant
10. Patients who received any investigational drug other than Tolvaptan within 30 days prior to the screening examination
11. Patients with general physical conditions, which may confound the results of the study, pose additional risk or preclude evaluation and assessments in this study

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2012-07; Primary Completion 2014-05 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Change in body weight at 4-day of treatment. | baseline and 4-day of treatment

SECONDARY OUTCOMES:
Change in Intake/Output Balance at 4-day of Treatment | baseline and 4-day of treatment
Change in Serum Sodium and Potassium Concentration at 4-day of treatment | baseline and 4-day of treatment
Treatment Failure at 4-day of Treatment | baseline and 4-day of treatment
Changes in Physician-assessed Signs and Symptoms of Heart Failure at 4-day of Treatment | baseline and 4-day of treatment
Changes in Patient Self-assessed Global Clinical Status at 4-day of Treatment | baseline and 4-day of treatment
Changes in Patient Self-assessed Dyspnea Status at 4-day of Treatment | baseline and 4-day of treatment
All-cause Mortality during the Study Period | Duration of hospital stay for 4 days, post-study follow up visit for 2 times
  Total timeframe expected average of 37 days for each participant

CONTACTS AND LOCATIONS:
Overall Officials: Chuen-Den Tseng, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospita, Taipei, Taiwan